CLINICAL TRIAL: NCT07212842
Title: METHYLENE BLUE-ENHANCED BLOOD WASHING DURING ZERO-BALANCE ULTRAFILTRATION REDUCES FLUID OVERLOAD AND INFLAMMATORY RESPONSE FOLLOWING CARDIOPULMONARY BYPASS: A RANDOMIZED CLINICAL TRIAL
Brief Title: Methylene Blue-Enhanced Ultrafiltration Improves Outcomes After Cardiopulmonary Bypass
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, André Timóteo Sapalo, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2.462.520
Record Dates: First submitted 2025-09-23; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Cardiopulmonary Bypass Surgery; Aortic Valve Surgery; Mitral Valve Surgery; Myocardial Revascularization Surgery With Extracorporeal Circulation
Keywords: Cardiac surgery; water overload; pulmonary congestion; intravascular volemia; cardiopulmonary bypass; zero-balance ultrafiltration; methylene blue
MeSH Terms: interventions — Methylene Blue

STUDY DESIGN:
Intervention Model Description: The objective of this study was to evaluate the effects of methylene blue blood lavage during zero-balance ultrafiltration (ZBUF) on fluid overload and the systemic inflammatory response. Patients were randomly assigned to one of three groups: conventional ultrafiltration (G-CUF; n = 43), saline blood lavage combined with ZBUF (G-ZBUF; n = 39), and methylene blue lavage combined with ZBUF (MB+G-ZBUF; n = 42). Fluid status was assessed using the InBody S10 precision bioimpedance device, which measured extracellular water (ECW), total body water (TBW), intracellular water (ICW), and the ECW/TBW ratio. Pulmonary congestion and intravascular volume were assessed separately with a Philips Lumify S4-1 transducer connected to a Samsung tablet. Pulmonary congestion was defined by the presence of B-lines on lung ultrasound. Intravascular volume was assessed using the inferior vena cava (IVC) distensibility index (DI) during mechanical ventilation and the collapsibility index (CI) during spontan
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional ultrafiltration (Active Comparator): Conventional ultrafiltration (G-CUF) patients in this group underwent conventional ultrafiltration widely used in cardiac surgery with extracorporeal circulation.
  Interventions: Drug: Methylene Blue; Procedure: Conventional ultrafiltration; Procedure: Zero-balance ultrafiltration
- Blood washing with physiological solution combined with zero-balance ultrafiltration (Placebo Comparator): Blood washing with physiological solution combined with zero-balanced ultrafiltration (G-ZBUF) patients in this group underwent zero-balanced ultrafiltration, and for this purpose, the simulation was performed with physiological solution.
  Interventions: Drug: Methylene Blue; Procedure: Conventional ultrafiltration; Procedure: Zero-balance ultrafiltration
- Methylene blue wash combined with zero-balanced ultrafiltration (Experimental): Methylene blue lavage combined with zero-balance ultrafiltration (MB+G-ZBUF). Patients assigned to this group underwent zero-balance ultrafiltration with concomitant blood lavage using methylene blue at a low dose of 1 mg/kg of body weight. Methylene blue was diluted in 1000 mL of 0.9% saline. An equivalent volume of fluid was simultaneously removed by zero-balance ultrafiltration, ensuring a balanced fluid state throughout the 20-minute procedure. For this purpose, a dedicated circuit was developed to allow simultaneous blood lavage and ultrafiltration. Blood was withdrawn through a dedicated port integrated into the SORIN oxygenator and directed by a centrifugal pump to a small reservoir containing the methylene blue solution. From this reservoir, the blood passed through a hemoconcentrator for filtration before being returned to the central reservoir of the cardiopulmonary bypass (CPB) circuit.
  Interventions: Drug: Methylene Blue; Procedure: Conventional ultrafiltration; Procedure: Zero-balance ultrafiltration

INTERVENTIONS:
Drug: Methylene Blue — This protocol was designed to perform intraoperative blood lavage with methylene blue at the end of surgery, with a duration of 20 minutes. A low dose of 1 mg/kg of body weight was administered. The objective was not to elicit hemodynamic effects, which require higher doses, but rather to exploit the anti-inflammatory and antioxidant properties of methylene blue.
  Methylene blue was diluted in 1000 mL of 0.9% saline. An equivalent volume of fluid was removed simultaneously by zero-balance ultrafiltration, maintaining a fluid-equilibrium state throughout the 20-minute procedure. For this purpose, a dedicated circuit was developed to enable concurrent blood lavage and ultrafiltration. Blood was withdrawn through a dedicated port integrated into the SORIN oxygenator and directed by a centrifugal pump to a small reservoir containing the methylene blue solution. From this reservoir, the blood passed through a hemoc
  Other Names: zero-balance ultrafiltration
Procedure: Conventional ultrafiltration — Conventional ultrafiltration (CUF). CUF during cardiopulmonary bypass (CPB) is performed to remove excess fluid and solutes from the patient's blood during cardiac surgery, thereby limiting fluid accumulation and attenuating pro-inflammatory effects. This technique increases hematocrit, improves cardiopulmonary function, and reduces the need for blood transfusions. Unlike modified ultrafiltration (MUF), which is performed after weaning from CPB, CUF is carried out simultaneously with CPB while the heart-lung machine remains in operation.
Procedure: Zero-balance ultrafiltration — Zero-balance ultrafiltration (Z-BUF). Z-BUF is performed during cardiopulmonary bypass (CPB) to maintain fluid equilibrium by removing plasma water and solutes while simultaneously infusing an equal volume of replacement fluid, thereby achieving a net zero fluid balance. This technique has been shown to decrease urine output, reduce tissue edema and the inflammatory response, improve arterial oxygenation (PaO₂), and lower the need for postoperative blood transfusions.

SUMMARY:
Introduction: Fluid overload and systemic inflammation are major contributors to postoperative complications in patients undergoing cardiac surgery with cardiopulmonary bypass (CPB). Objective: To evaluate the effects of blood washing with methylene blue during zero-balance ultrafiltration (ZBUF) on fluid overload and systemic inflammatory response. Methodology: Fluid status was assessed using the InBody S10 precision bioimpedance device, measuring extracellular water (ECW), total body water (TBW), intracellular water (ICW), and the ECW/TBW ratio. Pulmonary congestion and intravascular volume were evaluated separately using a Philips Lumify S4-1 transducer with a Samsung tablet. Pulmonary congestion was confirmed by the presence of B-lines on lung ultrasound. Intravascular volume was assessed via the inferior vena cava (IVC) distensibility index (DI) during mechanical ventilation and collapsibility index (CI) during spontaneous breathing. Inflammatory cytokine levels were measured using a Luminex xMAP-based multiplex immunoassay.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of cardiac disease requiring surgery with cardiopulmonary bypass (CPB)

Age ≥ 18 years

Ability to provide informed consent

Exclusion Criteria:

Chronic renal failure

Recent cardiac catheterization within the past month

Planned cardiac surgeries with an estimated CPB time of less than 60 minutes

Aortic surgery

Significantly impaired hepatic function

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2024-03-16 (Actual)

PRIMARY OUTCOMES:
Systemic Inflammation | Three years
  To assess systemic inflammation, blood samples were collected via central venous access through the internal jugular vein at five time points: before surgery, during surgery, 10 minutes after cannulation, 10 minutes after blood lavage with methylene blue and ultrafiltration, and 4 hours after ICU admission. Samples were drawn into EDTA-containing syringes (50 mM, pH 8.0) at one-tenth of the total blood volume. Plasma was separated by centrifugation at 1,700 × g for 10 minutes at 4 °C, transferred to new tubes avoiding the buffy coat, and centrifuged again at 11,000 × g for 2 minutes at 4 °C. Plasma was aliquoted and stored at -80 °C. Cytokine concentrations were quantified using a Luminex xMAP multiplex immunoassay (8-27-plex) in triplicate, enabling simultaneous measurement of up to seven cytokines, chemokines, and interleukins from 50 μL plasma.
Water overload | Three years
  Fluid balance was meticulously monitored, including fluids removed by conventional ultrafiltration, surgical suction, sponges, and urine output. Discrepancies between infused and removed volumes were corrected using zero-balance ultrafiltration (ZBUF), removing excess fluid or compensating deficits to match preoperative volemic status. For example, if 100 mL more than planned had been removed, only 900 mL were withdrawn. Body fluid composition was assessed with the InBody S10 bioimpedance device. Extracellular water (ECW) was measured at 5 kHz, total body water (TBW) at 250 kHz, and intracellular water (ICW) calculated as TBW-ECW. The ECW/TBW ratio served as the primary parameter to monitor fluid status and detect overload.
Intravascular volume assessment using IVC indices | Three years
  Intravascular volume will be evaluated by analyzing mechanical and hemodynamic changes in the inferior vena cava (IVC) using subcostal ultrasound images. The collapsibility index (CI = (IVCmax - IVCmin)/IVCmax) will be used during spontaneous breathing, and the distensibility index (DI = (IVCmax - IVCmin)/IVCmin) during mechanical ventilation.
  Time Frame: Preoperatively, immediately postoperatively, and 24 hours after surgery.
  Unit of Measure: Percentage (%).

SECONDARY OUTCOMES:
Length of stay in the intensive care unit (ICU) | Three years
  Secondary outcomes included the length of stay in the intensive care unit (ICU), measured in hours, to evaluate the clinical impact of zero-balance ultrafiltration with methylene blue. This parameter was recorded for all patients and analyzed in relation to fluid balance, pulmonary congestion, intravascular volume, and systemic inflammatory markers, providing a comprehensive assessment of the intervention's effects on postoperative recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo Medical School in Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No